CLINICAL TRIAL: NCT03577756
Title: Neurodevelopmental Assessment Outcomes of Infants With Cystic Fibrosis
Brief Title: Neurodevelopmental Assessment of Infants With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Akmer Mutlu, Associate professor, Hacettepe University
Other Study IDs: earlyrehabcysticfibrosis
Record Dates: First submitted 2018-06-23; First posted 2018-07-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Neurodevelopmental Disorders; Cystic Fibrosis
Keywords: cystic fibrosis; neurodevelopment; early rehabilitation
MeSH Terms: conditions — Neurodevelopmental Disorders; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with cystic fibrosis: Twelve months infants with cystic fibrosis will be assessed by the Bayley-III Baby and Child Development Assessment Scale (Bayley III) and the Rough Motor Function Measure.
  Interventions: Other: Neurodevelopmental assessments
- Healthy infants: Twelve months healthy infants will be assessed by the Bayley-III Baby and Child Development Assessment Scale (Bayley III) and the Rough Motor Function Measure.
  Interventions: Other: Neurodevelopmental assessments

INTERVENTIONS:
Other: Neurodevelopmental assessments — Infants' neurodevelopmental assessments will be done by the Bayley-III Baby and Child Development Assessment Scale (Bayley III) and the Gross Motor Function Measure. Bayley-III assess the development of five distinct scales to be consistent with areas of appropriate developmental assessment for children from birth to age 3. The Bayley-III revision includes Cognitive, Language, Motor, Social-Emotional, and Adaptive Behavior scales.The Gross Motor Function Measure (GMFM) has 5 dimensions: A-lying and roll- ing; B-sitting; C- kneeling and crawl- ing; D-standing; and E-walking, run- ning, and jumping. The items are scored from 0 to 3. All items are summarized and expressed as a value of total points for each dimension of the GMFM.

SUMMARY:
Infants included in the study will be divided into two groups as healthy infants and cystic fibrosis infants . Demographic, natal and postnatal information of the infants will be available from patient files. 12 months infants with cystic fibrosis and healthy infants will be assessed by the Bayley-III Baby and Child Development Assessment Scale (Bayley III) and the Gross Motor Function Measure. The assessment outcomes of healthy and cystic fibrosis infants will be compared.

ELIGIBILITY:
Inclusion Criteria:

* having diagnosis of cystic fibrosis
* to be postterm24-36 months old

Exclusion Criteria:

* Having congenital anomalies,
* Having an acute infection,
* Risk of high or low neurological impairment due to perinatal stroke, perinatal asphyxia, intra / peri-ventricular hemorrhage (IVH / PVL), bronchopulmonary dysplasia,
* The baby's family not reluctant to involved in study.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants with cystic fibrosis will be provided from the Hacettepe University Faculty of Medicine, Pediatric Chest Diseases Clinic and healthy infants will be provided from the Hacettepe University Department of Physiotherapy and Rehabilitation Developmental and Early Physiotherapy Unit.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure (GMFM) score | about 30 minutes
  It consists of a total of 88 items in the supine-posed position and during rotation, 17 items in sitting, 20 items in sitting, 14 items in crawling and kneeling, 13 items during standing, 24 items during walking-running-jumping. The child is scored according to the degree of achievement of gross motor functions in these materials. If the child can not initiate the activity 0 is given, can initiate independently 1 is given, can partially complete 2 is given, can independently complete 3 is given.
The Bayley Scales of Infant Development, Third Edition (BSID III) | about 30 minutes
  The Bayley-III includes Cognitive, Language, Motor, Social-Emotional, and Adaptive Behavior scales.
  Cognitive. The Cognitive scale of the Bayley-III contains 91 items. Language. This subtest contains 48 items. The Expressive Communication subtest assesses the individual's ability to vocalize, name pictures and objects, and communicate with others.
  Motor. The Bayley-III Motor scale include Fine Motor and Gross Motor subtests. The Fine Motor subtest contains 66 items and is purported to measure skills associated with eye movements, perceptual-motor integration, motor planning, and motor speed. The Gross Motor subtest contains 72 items and is designed to measure movements of the limbs and torso.
  Social-Emotional. This scale include 35 items, which measure emotional development and related behaviors.
  Adaptive Behavior. Bayley-III include the Adaptive Behavior Assessment System-Second Edition as a measure of adaptive skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sitrin MD, Lieberman F, Jensen WE, Noronha A, Milburn C, Addington W. Vitamin E deficiency and neurologic disease in adults with cystic fibrosis. Ann Intern Med. 1987 Jul;107(1):51-4. doi: 10.7326/0003-4819-107-1-51. PMID 3592448
- [Background] de Almeida Thomazinho P, de Miranda Chaves CR, Passaro CP, Meio MD. Motor delay in cystic fibrosis infants: an observational study. Early Hum Dev. 2011 Dec;87(12):769-73. doi: 10.1016/j.earlhumdev.2011.05.012. Epub 2011 Jun 15. PMID 21680118
- [Background] Singer L, Yamashita T, Lilien L, Collin M, Baley J. A longitudinal study of developmental outcome of infants with bronchopulmonary dysplasia and very low birth weight. Pediatrics. 1997 Dec;100(6):987-93. doi: 10.1542/peds.100.6.987. PMID 9374570
- [Derived] Tekerlek H, Yardimci-Lokmanoglu BN, Inal-Ince D, Ozcelik U, Mutlu A. Developmental Functioning Outcomes in Infants With Cystic Fibrosis: A 24- to 36-Month Follow-Up Study. Phys Ther. 2022 Jun 3;102(6):pzac037. doi: 10.1093/ptj/pzac037. PMID 35385120